CLINICAL TRIAL: NCT01370837
Title: Neurogenic Inflammation in Diabetic Polyneuropathy and Charcot Neuro-osteoarthropathy: Response to Intracutaneous Candida Albicans
Brief Title: Neurogenic Inflammation in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Dutch Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Kristy Pickwell, MD, Maastricht University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: METC 11-2-044
Record Dates: First submitted 2011-06-07; First posted 2011-06-10 (Estimated); Results first posted 2015-04-10 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes Mellitus; Polyneuropathies; Arthropathy, Neurogenic
MeSH Terms: conditions — Diabetes Mellitus; Polyneuropathies; Arthropathy, Neurogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy controls (Experimental)
  Interventions: Other: Intracutaneous injection of Candida albicans antigen.; Other: Temperature measurement.
- Diabetes (Experimental): Patients with diabetes mellitus without polyneuropathy.
  Interventions: Other: Intracutaneous injection of Candida albicans antigen.; Other: Temperature measurement.
- Polyneuropathy (Experimental): Patients with diabetes and polyneuropathy.
  Interventions: Other: Intracutaneous injection of Candida albicans antigen.; Other: Temperature measurement.

INTERVENTIONS:
Other: Intracutaneous injection of Candida albicans antigen. — Intracutaneous injection of 0.05 ml of four different concentrations of Candida albicans antigen on both the arm and foot.
Other: Temperature measurement. — Temperature measurement at the site of injection of the highest concentration of Candida albicans antigen on the foot and the same location on the contralateral foot using an infrared thermometer.

SUMMARY:
Polyneuropathy is a complication of diabetes mellitus which leads to decreased sensation in arms and legs. This in turn can lead to the development of (infected) foot ulcers. Charcot's disease can also be a consequence of polyneuropathy. Patients with Charcot's disease suddenly develop a red, warm and swollen foot, like an infection. Charcot's disease leads to foot fractures. After these fractures have healed, the shape of the foot can be dramatically altered. This altered shape of the foot increases the risk of developing foot ulcers. Nerves are important in regulating the inflammatory response. This study aims to investigate whether the inflammatory response is different in patients with polyneuropathy with and without a history of Charcot's disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes with and without polyneuropathy.
* Patients with type 2 diabetes with a history of Charcot's disease.
* Healthy controls.
* Signed informed consent.

Exclusion Criteria:

* Peripheral arterial disease: toe pressure < 70 mm Hg and/or transcutaneous oxygen tension < 40 mm Hg and/or claudication.
* Renal insufficiency: MDRD creatinin clearance < 30 ml/min.
* Systemic disease such as vasculitis or rheumatoid arthritis.
* Malignancy.
* (Diabetic) foot ulcer.
* Gout.
* Bacterial infection of an extremity.
* Skin condition of the dorsal aspect of the foot or the medial side of the upper arm.
* Bleeding disorder such as hemophilia.
* Use of medication for asthma.
* Impaired immunity such as in HIV/AIDS.
* Capillary blood glucose < 3 mmol/l or > 20 mmol/l at the time of the study.
* Peripheral oedema.
* Vaccination in the two months prior to study inclusion.
* Chemotherapy or radiation therapy in the twelve months prior to study inclusion.
* Surgery in the two months prior to study inclusion.
* Previous adverse reaction to Candida albicans antigen.
* Acute infection at the time of the study or in the month prior to study inclusion.
* Transfusion in the two months prior to study inclusion.
* Use of immunosuppressants in the two months prior to study inclusion.
* Pregnancy or breastfeeding.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas Schaper, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Pickwell K, Geerts M, van Moorsel D, Hilkman D, Kars M, Schaper NC. Regional differences in cell-mediated immunity in people with diabetic peripheral neuropathy. Diabet Med. 2020 Feb;37(2):350-355. doi: 10.1111/dme.14143. Epub 2019 Oct 10. PMID 31557355

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Controls | Diabetes | Polyneuropathy
Started | 12 | 12 | 17
Completed | 12 | 12 | 17
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Controls | Diabetes | Polyneuropathy | Total
Number analyzed (Participants) | 12 | 12 | 17 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (8.8) | 65 (6.7) | 66 (5.2) | 64 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 3 | 9
  Male | 8 | 10 | 14 | 32
Region of Enrollment [Number; unit: participants]
  Netherlands | 12 | 12 | 17 | 41

OUTCOME MEASURES:

1. Primary Outcome: Induration Size as a Response to Intracutaneous Candida Albicans.
Time Frame: 48 hours after injection.
Measure: Median (95% Confidence Interval); unit: millimeters
Arm/Group | Healthy Controls | Diabetes | Polyneuropathy
Number analyzed (Participants) | 12 | 12 | 17
millimeters
  Arm | 4 [1 to 13.5] | 6 [1.5 to 11] | 5 [2 to 6]
  Foot | 4 [0 to 9] | 2 [0 to 11.5] | 0 [0 to 1]
Statistical Analysis 1: Comparison: Healthy Controls vs Diabetes; Arm; Test type: Superiority or Other; p = 0.84, Kruskal-Wallis
Statistical Analysis 2: Comparison: Healthy Controls vs Diabetes; Foot; Test type: Superiority or Other; p = 0.76, Kruskal-Wallis
Statistical Analysis 3: Comparison: Diabetes vs Polyneuropathy; Arm; Test type: Superiority or Other; p = 0.53, Kruskal-Wallis
Statistical Analysis 4: Comparison: Diabetes vs Polyneuropathy; Foot; Test type: Superiority or Other; p = 0.07, Kruskal-Wallis
Statistical Analysis 5: Comparison: Healthy Controls; Arm vs foot; Test type: Superiority or Other; p = 0.25, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Diabetes; Arm vs foot; Test type: Superiority or Other; p = 0.27, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Polyneuropathy; Arm vs foot; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Healthy Controls | Diabetes | Polyneuropathy
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 1/17
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Controls (N=12) | Diabetes (N=12) | Polyneuropathy (N=17)
Allergic reaction to Candida antigen (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes